CLINICAL TRIAL: NCT02525367
Title: Clinical Pilot Study in the Feasibility and Effect of Online Cognitive Training on Cognitive Functions in Patients With Parkinson's Disease, Multiple Sclerosis and Depressive Patients Treated With Electroconvulsive Therapy
Brief Title: Online Cognitive Training in PD, MS and Depressed Patients Treated With Electroconvulsive Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: All Parkinson's disease patients have finished training. The MS and ECT groups have not finished as these groups had trouble including 20 patients.
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Parnassia Bavo Groep (Unknown); GGZ inGeest (Other)
Responsible Party: Principal Investigator, O.A. van den Heuvel, Mw. O.A. van den Heuvel, MD PhD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CWO/15-10E
Record Dates: First submitted 2015-08-06; First posted 2015-08-17 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Idiopathic Parkinson's Disease; Multiple Sclerosis; Elderly Post Electric Convulsive Therapy
Keywords: Parkinson's disease; Multiple Sclerosis; Depressed Elderly; Cognitive Dysfunction; Online Cognitive Training
MeSH Terms: conditions — Parkinson Disease; Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- PD-Experimental (Experimental): PD patients using the online cognitive training for 8 weeks, 3 times a week
  Interventions: Behavioral: Online cognitive training
- PD-Control (Active Comparator): PD patients using the active control condition for 8 weeks, 3 times a week
  Interventions: Behavioral: Active control condition
- MS-Experimental (Experimental): MS patients using the online cognitive training for 8 weeks, 3 times a week
  Interventions: Behavioral: Online cognitive training
- MS-Control (Active Comparator): MS patients using the active control condition for 8 weeks, 3 times a week
  Interventions: Behavioral: Active control condition
- postECT-Experimental (Experimental): Depressed elderly treated with ECT patients using the online cognitive training for 8 weeks, 3 times a week
  Interventions: Behavioral: Online cognitive training
- postECT-Control (Active Comparator): Depressed elderly treated with ECT patients using the active control condition for 8 weeks, 3 times a week
  Interventions: Behavioral: Active control condition

INTERVENTIONS:
Behavioral: Online cognitive training — The intervention is a computerized, online training programme which aims to train several cognitive abilities; especially the executive functions, attention, working memory and processing speed. The mental processes that are appealed to by the intervention are similar to processes that are trained in classic face-to-face training methods. Both the intervention protocol and the active control condition will contain several games that have the participant train cognitive functions/perform cognitive activities for 8 weeks, 3 times a week, 45-60 minutes each session.
  Other Names: BrainGymmer, Dezzel Media B.V., The Netherlands
  Arms: MS-Experimental; PD-Experimental; postECT-Experimental
Behavioral: Active control condition — The active control condition consists of cognitive activities that do not intend to train cognitive functions based on 'cristallized intelligence', such as trivia. Both the intervention protocol and the active control condition will contain several games that have the participant train cognitive functions/perform cognitive activities for 8 weeks, 3 times a week, 45-60 minutes each session.
  Arms: MS-Control; PD-Control; postECT-Control

SUMMARY:
In Parkinson's disease, Multiple Sclerosis and depressed patients treated with electroconvulsive therapy, cognitive dysfunction is prevalent. However, treatment of these dysfunctions is in its infancy.

The purpose of this study is 1) to assess the feasibility of a randomized controlled trial using an online computerized intervention for training cognitive abilities in the three patient groups and 2) to estimate the effect of the online training on objectively and subjectively measured cognitive functions.

The investigators hypothesize that patients using online cognitive training will improve more on cognitive functions, as compared to patients using an active control condition.

DETAILED DESCRIPTION:
In neurodegenerative disorders and psychiatric disorders, cognitive dysfunction is frequently reported. In Parkinson's disease (PD), Multiple Sclerosis (MS) and patients treated with electroconvulsive therapy after a severe or therapy resistant depression (postECT), executive dysfunction, attention deficit or episodic/autobiographic memory deficit is prevalent. In MS and PD, these dysfunctions can appear already early in the disease. The majority of PD patients - lifetime prevalence is about 80% - develops PD dementia. In MS, about half of the patients experiences problems with cognitive functions. ECT is used to treat patients with severe and/or therapy resistant depression. However, 30-50% of these patients develops severe cognitive dysfunction. Recovery usually occurs within six months after ECT. However, performances remain below-average compared to norm groups and there are large individual differences. The cognitive difficulties in MS and PD have a significant negative influence on the quality of life. Cognitive dysfunction in PD is associated with decreased independent daily functioning, hospitalization and the development and severity of neuropsychiatric symptoms. Furthermore, in the clinic cognitive dysfunction has been reported to be one of the most dreadful side effects of ECT. However, effective treatment of the described cognitive dysfunction is still in its infancy.

Cognitive training is based upon the principle that plasticity of the brain can facilitate function improvement by intensive training. In several neurological diseases, cognitive training has shown significant improvement in cognitive functions. In MS and PD, earlier studies have been small, frequently without an adequately controlled design. Additionally, earlier cognitive training programs have frequently been executed in a health care organization, impairing patients to successfully attend all training sessions due to mobility impairments. Also, there are limited studies in the effects of cognitive training on improved functioning of daily living and neuropsychiatric symptoms like anxiety and depression. Given the fact that there is an absence in cognitive training studies in patients post-ECT, there is no knowledge about the ability of cognitive training to speed up the natural course.

Using this pilot study, the investigators aim to study the feasibility of a randomized controlled trial using an online computerized intervention for training cognitive abilities in three patient groups. By using a double-blinded, controlled study design, the investigators keep in mind limitations of earlier comparable studies. If this treatment proves to be feasible, and a rough estimated effect size is positive, a larger randomized controlled trial can be executed to study the effectivity of this treatment. When effects are positive, an online cognitive training programme could prove to be a cost-efficient intervention that is accessible at home - something which is important for patients with mobility problems. The investigators hypothesize that patients using online cognitive training will improve more on cognitive functions, as compared to patients using an active training condition.

ELIGIBILITY:
Inclusion Criteria:

General criteria:

* Patients have (access to) a computer with access to the Internet. Patients are capable of using a keyboard and computer mouse.
* Patients are willing to sign informed consent.

PD-specific criteria:

* A compilation score of executive functions (i.e. Stroop, Trail Making Task, Fluency) shows deficit, which lies between 1 and 2 standard deviation (SD) below the mean of healthy Dutch norm population.
* Patients are diagnosed with Parkinson's disease according to the United Kingdom Parkinson's Disease Society Brain Bank criteria.
* Patients are in Hoehn & Yahr stadium < 4, and are medically stable during a month prior to the intervention. The medication will be attempted to remain stable for the remainder of the intervention.
* Patients are 50 to 70 years old.

MS-specific criteria:

* A compilation score of episodic memory (i.e. Rey Auditory Verbal Learning Test, Location Learning Test) shows deficit, which lies between 1 and 2 SD below the mean of healthy norm population.
* Patients have been diagnosed with MS for a period longer than three month prior to inclusion in this study according to the renewed McDonald criteria.
* Patients have been on stable medication for at least three months.
* Patients are 30 to 45 years old.

PostECT-specific criteria:

* Unipolar depressive patients indicated for ECT, who experience cognitive complaints after treatment with ECT.
* Patients have undergone the full ECT-procedure.
* Phonemic fluency and autobiographical memory (measured by the Kopelman Autobiographical Interview) show deficit: significant individual deterioration is present (> 1.5 SD deterioration), accounting for test- retest effects.
* Patients are 50 to 70 years old.

Exclusion Criteria:

General criteria:

* Indications for presence of dementia.
* Presence of traumatic brain injury.
* A psychiatric disorder (in the postECT group: other than unipolar depression).
* No history or presence of drug or alcohol abuse.
* Inability to undergo a neuropsychological assessment (e.g. due to fast fatigue, seeing problems or language barrier).

PD-specific criteria:

- Psychotic symptoms, as screened by the Questionnaire for Psychotic Experiences (QPE). Benign hallucinations with insight are not contraindicated).

MS-specific criteria:

- Patients with MS can't have relapses or can't use corticosteroids 4 weeks prior to the start of the study.

postECT-specific criteria:

- Indications for presence of delirium.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Feasibility | 8 weeks
  The feasibility of the intervention as reported by the patients on 4-point Likert scale items (T1)

SECONDARY OUTCOMES:
Trail Making Task | Baseline, 8 weeks and 12 weeks
  Cognitive functioning as assessed by neuropsychological measures. These are measured by the interaction effect between time of measurement (T0 versus T1, or T0 versus T2) and condition (experimental versus active control). If possible, parallel tests will be used to correct for repeated neuropsychological testing. The objectively measured intervention effect will be assessed on the most affected cognitive domain, different per syndrome:
  - PD and postECT: improvement in executive functions, measured by change in the Trail Making Task
Cognitive functioning (subjectively measured) | Baseline, 8 weeks and 12 weeks
  Change in subjective cognitive complaints as reported by the patient, measured by the Cognitive Failure Questionnaire (CFQ)
Feasibility | Patients will be interviewed in a group session after study completion, an expected average of half a year
  The feasibility of the intervention as reported by the patients in a group session lead by patients from the disease associations.
Stroop Color Word Task | Baseline, 8 weeks and 12 weeks
  Cognitive functioning as assessed by neuropsychological measures. These are measured by the interaction effect between time of measurement (T0 versus T1, or T0 versus T2) and condition (experimental versus active control). If possible, parallel tests will be used to correct for repeated neuropsychological testing. The objectively measured intervention effect will be assessed on the most affected cognitive domain, different per syndrome:
  - PD and postECT: improvement in executive functions, measured by change in the Stroop Color Word Test.
Letter Fluency | Baseline, 8 weeks and 12 weeks
  Cognitive functioning as assessed by neuropsychological measures. These are measured by the interaction effect between time of measurement (T0 versus T1, or T0 versus T2) and condition (experimental versus active control). If possible, parallel tests will be used to correct for repeated neuropsychological testing. The objectively measured intervention effect will be assessed on the most affected cognitive domain, different per syndrome:
  - PD and postECT: improvement in executive functions, measured by change in the Letter Fluency.
Rey Auditory Verbal Learning Test | Baseline, 8 weeks and 12 weeks
  Cognitive functioning as assessed by neuropsychological measures. These are measured by the interaction effect between time of measurement (T0 versus T1, or T0 versus T2) and condition (experimental versus active control). If possible, parallel tests will be used to correct for repeated neuropsychological testing. The objectively measured intervention effect will be assessed on the most affected cognitive domain, different per syndrome:
  - MS: improvement in episodic memory, measured by change in the Rey Auditory Verbal Learning Test.
Location Learning Test | Baseline, 8 weeks and 12 weeks
  Cognitive functioning as assessed by neuropsychological measures. These are measured by the interaction effect between time of measurement (T0 versus T1, or T0 versus T2) and condition (experimental versus active control). If possible, parallel tests will be used to correct for repeated neuropsychological testing. The objectively measured intervention effect will be assessed on the most affected cognitive domain, different per syndrome:
  - MS: improvement in episodic memory, measured by change in the Location Learning Test.

CONTACTS AND LOCATIONS:
Overall Officials: Odile A. Van den Heuvel, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc; Chris Vriend, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Background] Oudega ML, van Exel E, Wattjes MP, Comijs HC, Scheltens P, Barkhof F, Eikelenboom P, de Craen AJ, Beekman AT, Stek ML. White matter hyperintensities and cognitive impairment during electroconvulsive therapy in severely depressed elderly patients. Am J Geriatr Psychiatry. 2014 Feb;22(2):157-66. doi: 10.1016/j.jagp.2012.08.002. Epub 2013 Jan 11. PMID 23567440
- [Background] Chiaravalloti ND, DeLuca J. Cognitive impairment in multiple sclerosis. Lancet Neurol. 2008 Dec;7(12):1139-51. doi: 10.1016/S1474-4422(08)70259-X. PMID 19007738
- [Background] Bosboom JL, Stoffers D, Wolters ECh. Cognitive dysfunction and dementia in Parkinson's disease. J Neural Transm (Vienna). 2004 Oct;111(10-11):1303-15. doi: 10.1007/s00702-004-0168-1. Epub 2004 Jun 30. PMID 15480840
- [Background] Rubin EH, Kinscherf DA, Figiel GS, Zorumski CF. The nature and time course of cognitive side effects during electroconvulsive therapy in the elderly. J Geriatr Psychiatry Neurol. 1993 Apr-Jun;6(2):78-83. doi: 10.1177/089198879300600204. PMID 8512634
- [Background] Achiron A, Barak Y. Cognitive impairment in probable multiple sclerosis. J Neurol Neurosurg Psychiatry. 2003 Apr;74(4):443-6. doi: 10.1136/jnnp.74.4.443. PMID 12640060
- [Background] Muslimovic D, Post B, Speelman JD, Schmand B. Cognitive profile of patients with newly diagnosed Parkinson disease. Neurology. 2005 Oct 25;65(8):1239-45. doi: 10.1212/01.wnl.0000180516.69442.95. PMID 16247051
- [Background] Aarsland D, Andersen K, Larsen JP, Lolk A, Kragh-Sorensen P. Prevalence and characteristics of dementia in Parkinson disease: an 8-year prospective study. Arch Neurol. 2003 Mar;60(3):387-92. doi: 10.1001/archneur.60.3.387. PMID 12633150
- [Background] Hely MA, Reid WG, Adena MA, Halliday GM, Morris JG. The Sydney multicenter study of Parkinson's disease: the inevitability of dementia at 20 years. Mov Disord. 2008 Apr 30;23(6):837-44. doi: 10.1002/mds.21956. PMID 18307261
- [Background] Rao SM, Leo GJ, Bernardin L, Unverzagt F. Cognitive dysfunction in multiple sclerosis. I. Frequency, patterns, and prediction. Neurology. 1991 May;41(5):685-91. doi: 10.1212/wnl.41.5.685. PMID 2027484
- [Background] Klepac N, Trkulja V, Relja M, Babic T. Is quality of life in non-demented Parkinson's disease patients related to cognitive performance? A clinic-based cross-sectional study. Eur J Neurol. 2008 Feb;15(2):128-33. doi: 10.1111/j.1468-1331.2007.02011.x. PMID 18217883
- [Background] Fletcher P, Leake A, Marion MH. Patients with Parkinson's disease dementia stay in the hospital twice as long as those without dementia. Mov Disord. 2011 Apr;26(5):919. doi: 10.1002/mds.23573. Epub 2011 Mar 21. No abstract available. PMID 21425337
- [Background] Cicerone KD, Langenbahn DM, Braden C, Malec JF, Kalmar K, Fraas M, Felicetti T, Laatsch L, Harley JP, Bergquist T, Azulay J, Cantor J, Ashman T. Evidence-based cognitive rehabilitation: updated review of the literature from 2003 through 2008. Arch Phys Med Rehabil. 2011 Apr;92(4):519-30. doi: 10.1016/j.apmr.2010.11.015. PMID 21440699
- [Background] Olazaran J, Reisberg B, Clare L, Cruz I, Pena-Casanova J, Del Ser T, Woods B, Beck C, Auer S, Lai C, Spector A, Fazio S, Bond J, Kivipelto M, Brodaty H, Rojo JM, Collins H, Teri L, Mittelman M, Orrell M, Feldman HH, Muniz R. Nonpharmacological therapies in Alzheimer's disease: a systematic review of efficacy. Dement Geriatr Cogn Disord. 2010;30(2):161-78. doi: 10.1159/000316119. Epub 2010 Sep 10. PMID 20838046
- [Background] Hindle JV, Petrelli A, Clare L, Kalbe E. Nonpharmacological enhancement of cognitive function in Parkinson's disease: a systematic review. Mov Disord. 2013 Jul;28(8):1034-49. doi: 10.1002/mds.25377. Epub 2013 Feb 20. PMID 23426759
- [Background] Rosti-Otajarvi EM, Hamalainen PI. Neuropsychological rehabilitation for multiple sclerosis. Cochrane Database Syst Rev. 2011 Nov 9;(11):CD009131. doi: 10.1002/14651858.CD009131.pub2. PMID 22071863
- [Background] Hughes AJ, Daniel SE, Kilford L, Lees AJ. Accuracy of clinical diagnosis of idiopathic Parkinson's disease: a clinico-pathological study of 100 cases. J Neurol Neurosurg Psychiatry. 1992 Mar;55(3):181-4. doi: 10.1136/jnnp.55.3.181. PMID 1564476
- [Background] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374